CLINICAL TRIAL: NCT03198468
Title: Vapor Ablation for Localized Cancer Lesions of the Lung - A Clinical Feasibility Treat-and Resect Study (VAPORIZE)
Brief Title: Vapor Ablation for Localized Cancer Lesions of the Lung (VAPORIZE)
Acronym: VAPORIZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uptake Medical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-2402
Record Dates: First submitted 2017-06-14; First posted 2017-06-26 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Non Small Cell Lung Cancer; Metastatic Lung Cancer; Lung Cancer
Keywords: Non Small Cell Lung Cancer; Metastatic Lung Cancer; Lung Cancer; Vapor Ablation; BTVA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vapor Ablation (Experimental)
  Interventions: Device: Bronchoscopic Thermal Vapor Ablation

INTERVENTIONS:
Device: Bronchoscopic Thermal Vapor Ablation — Vapor (steam) is infused into the targeted region for 8 seconds at a precisely controlled flow rate and power (an energy level of 330 calories).

SUMMARY:
This study is a prospective, single-arm, multi-center, pilot trial of Bronchoscopic Thermal Vapor Ablation for Lung Cancer (BTVA-C) in patients with primary lung cancer or metastatic cancer in the lung. Patients who have consented to participate in this study (enrolled) will be subject to eligibility screening and baseline assessments, prior to undergoing the BTVA-C procedure. Only patients that meet all of inclusion criteria and none of the exclusion criteria will receive vapor ablation treatment.

Patients will receive BTVA-C treatment followed by standard-of-practice surgical resection.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, multi-center, pilot trial of Bronchoscopic Thermal Vapor Ablation for Lung Cancer (BTVA-C) in patients with primary lung cancer or metastatic cancer in the lung.

Subjects identified for this study will be those that have a surgical resection already scheduled as part of their lung cancer treatment. Patients who have consented to participate in this study (enrolled) will undergo screening assessments to evaluate the inclusion criteria associated with their lung cancer and general health. Only patients that meet all of the inclusion criteria and none of the exclusion criteria will be scheduled for treatment with the BTVA-C System.

A total of 8 subjects will be treated at up to 2 investigational sites in Australia.

Prior to the vapor ablation procedure, the patient's CT scan is analyzed to evaluate the location and size of the target lesion. The segments and airways associated with the lesion are identified and images are created to aid in the navigation to appropriate treatment locations during the upcoming procedure.

At the time of the vapor ablation procedure, the Uptake catheter is placed in a selected airway with a thin bronchoscope. A balloon at the distal end of the catheter is then inflated to occlude the bronchus prior to vapor infusion. Sterile water is heated to approximately 100°-140°C by a reusable Generator and vapor (steam) is infused into the targeted region for 8 seconds at a precisely controlled flow rate and power. If necessary, the catheter is moved to the next airway and the procedure is repeated until all desired airways have been treated (maximum 3 treatments). The treatment creates a uniform field of necrosis in the parenchyma around the lesion.

The interval between vapor ablation and the surgical resection will be a minimum of 60 hours to a maximum of 105 hours, with the exact scheduling determined by the investigator. The resected tissue will undergo pathological evaluation for tissue viability.

In addition to standard post-operative follow-up, patients will be evaluated at Day 7 (± 2 days) and Day 30 (± 5 days) post-resection to assess safety and feasibility.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old
2. Non-small cell lung cancer tumor(s) ≤ 2cm (T1aN0, T1bN0, T1aN1, or T1bN1) suitable for resection OR Metastatic lung tumor(s) ≤ 2cm suitable for resection
3. Suitable candidate for resection per standard of practice
4. Microscopic proof of malignancy obtained.
5. Location of tumor:

   1. In periphery of lung (outermost 1/3)
   2. Anticipation that resection would remove all gross tumor and ablation with grossly negative margins
   3. Maximum of three vapor ablation applications would target entire margin according to the vapor ablation plan
6. Signed informed consent

Exclusion Criteria:

1. Centralized tumor not amenable to resection (abutting main stem bronchus, main pulmonary artery branches, esophagus, or trachea)
2. Carcinoid lung tumors
3. Tumor is associated with atelectasis or obstructive pneumonitis or pleural effusion
4. Pulmonary function tests (PFTs): post-bronchodilator forced expired volume in one second (FEV1) or forced vital capacity (FVC) < 50% predicted, diffusing capacity of the lung for carbon monoxide (DLCO) <50% predicted
5. Requirement for supplemental oxygen at rest or exercise
6. Hospitalization for cardiac disease within the preceding 6 months
7. Liver enzymes (ALP, ALT, AST) or total bilirubin > 1.5 upper limit of normal (ULN)
8. Serum creatinine > 2 mg/dl
9. Recent infection (within 30 days)
10. Receiving immunosuppressive medication or prednisone > 10 mg/day (or equivalent)
11. Pre-existing implants within the airways that impede navigation to the target lesion
12. Pregnant or breastfeeding women and those of childbearing potential who are not practicing a reliable form of contraception
13. Disorder of coagulation, history of severe hemoptysis, or receiving anticoagulant medication. Antiplatelet medication is permitted provided that the medication can be held a minimum of 7 days prior to the procedure and 10 days, post-procedure.
14. Any condition that in the opinion of the investigator or reviewer may interfere with the safety of the patient or evaluation of the study objectives
15. Any tumor characteristic that in the opinion of the investigator or reviewers may interfere with the safety of the patient or evaluation of the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
AEs and SAEs related to BTVA-C procedure | Day 30 follow-up
  The number of reported adverse events (AEs), serious adverse events (SAEs) related to the BTVA-C procedure.
Successful BTVA-C Treatment Delivery | 1 day post-ablation
  Treatment meets 100% of the required procedural steps/requirements per the Instructions For Use (IFU) and treatment is delivered to the target tumor per the individual patient navigational plan
Ischemic tissue assessment | 2-4 days post-ablation (pre surgical resection)
  CT Imaging to identify and assess ischemic tissue
Tissue necrosis evaluated by semi-quantitative histological analysis | 1 day post-surgical resection
  Semi-quantitative scoring of necrotic tissue assessed by histology

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Steinfort, MD, PhD, Principal Investigator — Melbourne Health, The Royal Melbourne Hospital, City Campus.
Locations (1):
- The Royal Melbourne Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Uptake Medical Website — http://www.uptakemedical.com/